CLINICAL TRIAL: NCT06286605
Title: Horizontal Ridge Augmentation Using One-stage Guided Bone Regeneration (GBR) for Bone Defect Class IV of Cawed and Howell With Collagene Membrane (OssMem) and a Mix of Bovine Bone Substitute (A-Oss) and Autogenous Bone Versus A-Oss and LCR-A, a Synthetic Bone : a Randomized Controlled Trial
Brief Title: RCT GBR One Stages Comparing A-Oss and Autogenous Bone Versus A-Oss and LCR-A
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi di Sassari (Other)
Collaborators: Melodia, Dario, M.D. (Individual); Pisano, Milena, M.D. (Individual); Dr. Aurea Lumbau (Unknown); Prof. Silvio Mario Meloni (Unknown); Prof. Edoardo Baldoni (Unknown)
Responsible Party: Principal Investigator, Marco Tallarico, Aisstent Professor, Università degli Studi di Sassari
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UNISS_PHD_Osstem_4
Record Dates: First submitted 2023-04-24; First posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Guided Bone Regeneration; Dental Implant
Keywords: Dental Implant; GBR

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized controlled trial of parallel-group design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A-oss and autogenous bone (Experimental): In these group a GBR will be performed using only A-oss and autologous bone will be added and then will be covered with a membrane.
  Interventions: Procedure: A-oss and autogenous bone
- A-oss and LCR-A (Active Comparator): In these subjects a GBR will be performed using only A-oss and LCR-A and then will be covered with a membrane.
  Interventions: Procedure: A-oss an LCR-A

INTERVENTIONS:
Procedure: A-oss and autogenous bone — Horizontal ridge augmentation in one stages approach will be performed using a mix of A-Oss and autologenous bone.
  Arms: A-oss and autogenous bone
Procedure: A-oss an LCR-A — Horizontal ridge augmentation in one stages approach will be performed using OssMem with A-Oss and LCR-A
  Arms: A-oss and LCR-A

SUMMARY:
The aim of this randomized controlled trial is to evaluate the tridimensional bone stability after horizontal one-stage GBR using collagene membrane (OssMem) with a mix of Bovine Bone Substitute (A-Oss) and autogenous bone (test group) versus A-Oss and LCR-A, a synthetic bone (control group).

ELIGIBILITY:
Inclusion Criteria:

* Patients that required an implant supported restoration and staged horizontal guided bone regeneration (defect of class IV according to Cawed and Howell) in both mandible or maxilla.
* Patents able to understand and sign an informed consent.
* Patients were to be 18 years or older with a residual horizontal ridge thickness of 4 mm or less (Cawood-Howell Class III- IV) in the intended implant site.
* Smokers will be categorized into: 1) non smokers; 2) moderate smokers (smoking up to 10 cigarettes/day); 3) heavy smokers (smoking more than 11 cigarettes/day). Only categories 1 and 2 will be included.

Exclusion Criteria:

* General contraindications to implant surgery.
* Patients irradiated in the head and neck area.
* Immunosuppressed or immunocompromised patients.
* Patients treated or under treatment with intravenous amino-bisphosphonates.
* Patients with untreated periodontitis.
* Patients with poor oral hygiene and motivation.
* Uncontrolled diabetes.
* Pregnancy or nursing.
* Substance abuser.
* Heavy smokers (smoking more than 11 cigarettes/day).
* Psychiatric problems or unrealistic expectations.
* Lack of opposite occluding dentition in the area intended for implant placement.
* Immediate implants (extractive sites will have to be healed from 6-8 weeks).
* Patients participating in other studies, if the present protocol cannot be properly adhered to.
* Patients referred only for implant placement and cannot be followed ant the treating centre.
* Patients unable to be followed for 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Rate of Implants survival | Up to 5 years
  Defined as implant mobility and/or any infection dictating implant removal, and/or implant fracture and/or any other mechanical complication rendering the implant unusable. The stability of each individual implant will be measured by the local blinded outcome assessors manually tightening the screws with a torque of 30 Ncm at abutment connection at initial loading. At 1,3 and 5 years after loading, individual implants will be manually tested for stability. Once the single crowns will be screwed, their stability will be assessed by rocking the crown with the handles of two dental instruments
Number of Participants with prosthesis failure | Up to 5 years
  Whether it will not be possible to place the prosthesis because of implant failure or a prosthesis that has to be remade for any reason.
Number of complications | Up to 5 years
  Technical (fracture of the framework and/or the veneering material, screw loosening, etc.) and/or biologic (pain, swelling, mobility, membrane exposure, suppuration) complications will be considered

SECONDARY OUTCOMES:
Horizontal and volumetric dimensional changes | 6 and 12 months
  CBCT scans will perform before ridge reconstruction and six months after. The Digital Imaging and Communication in Medicine (DICOM) data will export the OnDemand 3D software version 1.0.9.3223 (Cybermed Inc., Seoul, Korea) to perform all measurements. The DICOM data were manually alined basic on unchanged anatomical areas (e.g., teeth, basal skull, implants) and then automatically matched using the Fusion adjunctive module (Cybermed Inc. Seoul, Korea). Horizontal bone measure will recorded for all reconstructed ridge 2 mm below the bone crest, before and after treatment. Then, the postoperative volumetric data were subtracted to the original scenario. The new generated set of DICOM data will stored as a separately files. Volumetric measurements of grafts were performed with OnDemand 3D software (Cybermed Inc., Seoul, Korea) using the previously generated set of DICOM data.The volumes of the grafted material will calculated using automatic tools, basing on its opacity.
Rate of peri-implant marginal bone level | At 1,3 and 5 years
  Peri-implant marginal bone level changes will be assessed on periapical radiographs took with the paralleling technique at implant placement, at initial loading, 1,3 and 5 years after loading. Ideally digital radiographs should be taken, otherwise radiographs on conventional films will be scanned into TIFF format with a 600 dpi resolution, and stored in a personal computer. Peri-implant marginal bone levels will be measured using the Scion Image (Scion Corporation, Frederick, MD, USA) software. The software will be calibrated for every single image using the known distance of the first two consecutive threads. Measurements of the mesial and distal bone crest level adjacent to each implant will be made to the nearest 0.01 mm. Reference points for the linear measurements will be: the coronal margin of the implant collar and the most coronal point of bone-to-implant contact. Bone levels will be measured.
Plaque Index and bleeping on probing | At 1,3 and 5 years
  Plaque index (PI), defined as plaque absent or present (0/1), and Bleeding on Probing (BoP), defined as bleeding on probing absent or present (0/1), will recorded 1,3 and 5 years after final prosthesis delivery. One assessor, not previously involved in the study, made all the clinical outcomes.
Valuation of patient satisfaction | At 1,3 and 5 years
  Patients will answer the following questions (separately for each implant):
  1. Are you satisfied with the function of your implant-supported prostheses? Possible answers: yes absolutely, yes partly, not sure, not really, absolutely not.
  2. Are you satisfied with the aesthetic outcome of your implant-supported prostheses? Possible answers: yes absolutely, yes partly, not sure, not really, absolutely not.
  3. Would you undergo the same therapy again? Possible answers: "yes" or "no".1) Are you satisfied with the function of your implant-supported prostheses? Possible answers: yes absolutely, yes partly, not sure, not really, absolutely not.
  2) Are you satisfied with the aesthetic outcome of your implant-supported prostheses? Possible answers: yes absolutely, yes partly, not sure, not really, absolutely not.
  3) Would you undergo the same therapy again? Possible answers: "yes" or "no".
Valuation of soft tissue thickness and amount of keratinized tissue | At 1,3 and 5 years
  The soft tissue biotype will be investigated by the same surgeon at the surgical procedures using a periodontal probe into the sulcus. Greater will be the thickness of the tissue, smaller will be transparency of the periodontal probe. The amount of keratinized tissue will be evaluated 1 year after surgical procedures using a periodontal probe. This outcome will be evaluated according to the distance from the gingival margin to the mucogingival junction
Rate of pes score | At 1,3 and 5 years
  Esthetic evaluation of occlusal and vestibular pictures will take every years after definite loading was done following the pink esthetic score (PES). In brief, the PES score evaluates seven variables: mesial papilla, distal papilla, soft tissue level, soft tissue contour, alveolar process deficiencies, soft tissue color and texture. A 0-1-2 scoring system was used, 0 being the lowest and 2 being the highest value, with a maximum achievable score of 14 per dental unit.

CONTACTS AND LOCATIONS:
Locations (1):
- Marco Tallarico, Sassari, Italy

IPD SHARING:
Plan to Share IPD: No